CLINICAL TRIAL: NCT00833794
Title: A Two-Arm Study Comparing the Analgesic Efficacy and Safety of Tramadol HCl Once-a-Day Versus Placebo for the Treatment of Pain Due to Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT3-005; NCT00833794 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2009-08-10 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Pain; Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 Tramadol Once A Day (Experimental)
  Interventions: Drug: Tramadol Once a day
- 2 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol Once a day
  Arms: 1 Tramadol Once A Day
Drug: Placebo
  Arms: 2 Placebo

SUMMARY:
The purpose of this study is to compare the analgesic efficacy, safety and clinical benefit of Tramadol OAD tablets versus Placebo.

ELIGIBILITY:
Inclusion Criteria for Open-Label phase:

1. Males or females
2. Must be between the ages of 40-80
3. Must meet the American College of Rheumatology (ACR) Clinical Classification Criteria for Osteoarthritis of the Knee:

   * Current knee pain
   * Less than 30 minutes of morning stiffness with or without crepitus on active motion
   * Confirmation either by arthroscopy or radiologist's report (X-rays showing osteophytes, joint space narrowing or subchondral bone sclerosis {eburnation}) within five years prior to entry into the study
4. Must have a history of exposure to treatment (for pain due to osteoarthritis (OA) of the knee) with Non-steroidal anti-inflammatory drugs (NSAIDs), COX II inhibitors or tramadol.
5. Must be taking one of the above medications on a regular basis in the 30 days prior to Visit 2 (S0).
6. Must meet the following criteria for severity of pain at Visit 2 (Day S0):

   * Have a score of ≥ 4 on the 11-point Numerical Rating Scale (PI-NRS; range: 0-10)
   * Have a total increase of ≥ 2 points on the 11-point Numerical Rating Scale (range: 0-10) compared to the rating at Visit 1 (Day SX)
7. Must have a erythrocyte sedimentation rate (ESR) < 40 mm/hr
8. Must have oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials
9. Must have signed and dated an approved written Informed Consent form in French, Spanish, English or Romanian, which has also been signed and dated by the Investigator (unless otherwise required by the ethics committee), prior to study participation

Exclusion Criteria for Open-Label phase:

1. Has known rheumatoid arthritis or any other rheumatic disease
2. Has secondary arthritis i.e. any of the following: septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; target joint fracture; acromegaly; fibromyalgia; Wilson's disease; Ochronosis; Haemochromatosis; Osteochondromatosis; heritable arthritic disorders; or collagen gene mutations
3. Has a history of bursitis of the knee (target knee)
4. Has a history of pain in the ipsilateral hip (target knee)
5. Has had a meniscal tear in the target knee within the last 12 months
6. Has had cartilage reconstruction procedure in the target knee
7. Has had a therapeutic arthroscopy procedure in the target knee within the last 12 months
8. Has a Body Mass Index (BMI) greater than 37
9. Has had a major illness, requiring hospitalisation during the 3 months before commencement of the screening period
10. Is unwilling to stop taking pain medication other than the study medication (for arthritis or other types of pain) or is unwilling to stop taking other medications for the treatment of OA
11. Has previously failed treatment with tramadol or discontinued treatment with tramadol due to adverse events
12. Has been taking other opioids (e.g. codeine, oxycodone, hydromorphone, etc.) for treatment of OA or other chronic conditions
13. Has received Corticosteroid Injections in the target knee within the last 3 months or Viscous injections in the target knee within the last 6 months
14. Has had treatment within the last 3 weeks with any of the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors; serotonin-norepinephrine reuptake inhibitors or any other drug that reduces seizure threshold
15. Has had treatment with another investigational agent within the last 30 days
16. Has a history of seizure disorder other than Infantile Febrile Seizures
17. Has a previous or current opioid dependency
18. Has a bowel disease causing malabsorption
19. Is pregnant, lactating or of childbearing potential and is unwilling to utilise a medically approved method of contraception during participation in this clinical trial
20. Has significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range
21. Has significant renal disease (defined as creatinine clearance <30 mL/min
22. Has a history of current or past substance abuse or dependence, other than nicotine
23. Has a known and documented allergy to tramadol or any structurally similar drugs (e.g. opiates)
24. Has a known and documented allergy to acetaminophen or any structurally similar drugs
25. Has any other condition that, in the opinion of the Investigators, would adversely affect the patient's ability to complete the study or its measures.

Inclusion criteria for the double-blinded phase:

* Patients must continue to meet the open-label eligibility criteria and
* Must have a score of ≥ 4 on the Numerical Rating Scale (NRS) with a total increase of ≥ 2 points on the NRS compared to Visit 3(Day R14) and
* Must not have taken any of the prohibited medications during the Open-label Phase.

Exclusion criteria for the double-blinded phase:

* Patient Request
* Adverse Events that contraindicate further administration of the study medication
* Any other situation where in the opinion of the Investigator continued participation in the study would not be in the patient's best interest.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2004-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

REFERENCES:
- [Result] Burch F, Fishman R, Messina N, Corser B, Radulescu F, Sarbu A, Craciun-Nicodin MM, Chiriac R, Beaulieu A, Rodrigues J, Beignot-Devalmont P, Duplan A, Robertson S, Fortier L, Bouchard S. A comparison of the analgesic efficacy of Tramadol Contramid OAD versus placebo in patients with pain due to osteoarthritis. J Pain Symptom Manage. 2007 Sep;34(3):328-38. doi: 10.1016/j.jpainsymman.2006.11.017. Epub 2007 Jun 21. PMID 17583466
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Period: Open-label Phase
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Started | 1028 (Enrolled. Population described in the baseline characteristics is 1023 patients (Open-Label safety).) | 0 (No Placebo arm during open-label phase.)
Entered run-in Period | 1027 | 0
Received Open-Label Treatment | 1023 | 0
Completed | 646 (Randomized in double-blind phase) | 0
Not Completed | 382 | 0
Not completed — Adverse Event | 225 | 0
Not completed — Lack of Efficacy | 28 | 0
Not completed — Withdrawal by Subject | 48 | 0
Not completed — Physician Decision | 20 | 0
Not completed — Administrative reason | 1 | 0
Not completed — Protocol Violation | 47 | 0
Not completed — Did not complete wash-out period | 12 | 0
Not completed — enrolled in error (immediately D/C) | 1 | 0
Period: Double-blind Phase
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Started | 432 (Of the 646 patients who completed the Open-Label phase, 432 were randomized to Tramadol Once A Day) | 214 (Of the 646 patients who completed the Open-Label phase, 214 were randomized to Placebo)
Completed | 326 | 165
Not Completed | 106 | 49
Not completed — Adverse Event | 44 | 11
Not completed — Lack of Efficacy | 34 | 22
Not completed — Withdrawal by Subject | 23 | 6
Not completed — Physician Decision | 4 | 7
Not completed — Administrative reason | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Tramadol Once A Day | 2 Placebo | Total
Number analyzed (Participants) | 432 | 214 | 646
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 116 | 368
  >=65 years | 180 | 98 | 278
Age Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0) | 62.3 (8.9) | 62.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 133 | 408
  Male | 157 | 81 | 238

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score as Measured by the 11-point Pain Intensity-Numerical Rating Scale Score at the End of the Study (Week 12 or Time of Discontinuation)
Description: The Pain Intensity Score is an 11-point pain intensity numerical rating scale ranging from 0: no pain to 10: worst possible pain. The mean score at the end of the study (week 12 or time of discontinuation) was calculated.
Time Frame: 12 weeks
Population: Full analysis population: all randomized patients who received at least one dose of the randomized study medication regardless of the status of the post-dosing assessment.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
Points on a scale | 4.3 (2.5) | 4.8 (2.4)

2. Secondary Outcome: Pain Intensity Score (11-point PINRS) After 6 Weeks of Maintenance Treatment
Description: The Pain Intensity Score is an 11-point pain intensity numerical rating scale ranging from 0: no pain to 10: worst possible pain
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
Points on a scale | 4.0 (2.2) | 4.5 (2.2)

3. Secondary Outcome: Pain Intensity Score Stratified by Dose, at the End of the Study (Week 12 or Time of Discontinuation)
Description: Pain Intensity Score (an 11-point pain intensity numerical rating scale ranging from 0: no pain to 10: worst possible pain) was stratified by final dose level, at week 12 or time of discontinuation. The final optimum dose level based upon efficacy and tolerability was kept for the entire study. The mean score was calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 1 Tramadol Once A Day | 2 Placebo | Tramadol Once A Day 200 mg | Tramadol Once A Day 300 mg
Number analyzed (Participants) | 431 | 214 | 106 | 325
Points on a scale | 4.3 (2.5) | 4.8 (2.4) | 4.1 (2.4) | 4.4 (2.6)

4. Secondary Outcome: WOMAC Pain Subscale Score at the End of the Study (Week 12 or Time of Discontinuation)
Description: Mean WOMAC Pain Subscale score at week 12. The WOMAC scale is a 24-item questionnaire divided in 3 subscales, using a 5-point Likert-scale ranging from no difficulty to extreme difficulty (0-none; 1-slight; 2-moderate; 3-severe; 4-extreme). The WOMAC pain subscale results from the sum of 5 pain questions. The maximum total score is 20.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
Points on a scale | 6.9 (4.0) | 7.5 (4.1)

5. Secondary Outcome: WOMAC Physical Function Subscale Score at the End of the Study (Week 12 or Time of Discontinuation)
Description: Mean WOMAC Physical Function Subscale score at week 12. The WOMAC scale is a 24-item questionnaire divided in 3 subscales, using a 5-point Likert-scale ranging from no difficulty to extreme difficulty (0-none; 1-slight; 2-moderate; 3-severe; 4-extreme). The WOMAC Physical Function subscale results from the sum of 17 physical function questions and the maximum possible score is 68.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
Points on a scale | 24.9 (13.4) | 27.5 (13.8)

6. Secondary Outcome: Patient Global Impression of Change at the End of the Study (Week 12 or Time of Discontinuation)
Description: This assessment of overall status integrates the effect of the treatment on pain, side effects, and the patient's expectation of pain relief. It is made using a 7-point categorical scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 425 | 210
participants
  1 = very much improved | 86 | 27
  2 = much improved | 148 | 59
  3 = minimally improved | 108 | 58
  4 = no change | 49 | 42
  5 = minimally worse | 17 | 13
  6 = much worse | 17 | 8
  7 = very much worse | 0 | 3

7. Secondary Outcome: Physician Global Impression of Change at the End of the Study (Week 12 or Time of Discontinuation)
Description: This assessment of overall impression of study drug is made using a 7-point categorical scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse)
Time Frame: week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 423 | 210
participants
  1 = very much improved | 76 | 25
  2 = much improved | 154 | 71
  3 = minimally improved | 108 | 49
  4 = no change | 49 | 41
  5 = minimally worse | 21 | 17
  6 = much worse | 13 | 5
  7 = very much worse | 1 | 2
  Not determined | 1 | 0

8. Secondary Outcome: Time to Response
Description: Response was defined as a decrease of ≥1 point in an 11-point PINRS (11-point pain intensity numerical rating scale ranging from 0: no pain to 10: worst possible pain) from baseline to the last visit. The time to response was estimated using Kaplan-Meier analysis and a 95% CI for the median time was calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
days
  1-point response | 14 [14 to 14] | 14 [14 to 14]
  2-point response | 14 [14 to 15] | 15 [14 to 16]
  3-point response | 16 [15 to 35] | 39 [35 to 56]
  4-point response | 15 [14 to 15] | 35 [35 to 56]
  5-point response | 35 [15 to 35] | 77 [56 to 99]

9. Secondary Outcome: Discontinuation Due to Lack of Efficacy
Description: The number of patients who discontinued due to lack of efficacy was reported.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
participants | 34 | 22

10. Secondary Outcome: Discontinuation Due to Adverse Events
Description: The number of patients who discontinued due to adverse events (AEs). An AE is defined as any untoward medical event that occurs during the course of a clinical investigation in which a patient is administered a pharmaceutical or other therapeutic product. Its occurrence does not necessarily imply a causal relationship with the treatment.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Number analyzed (Participants) | 431 | 214
participants | 44 | 12

ADVERSE EVENTS:
Arm/Group | 1 Tramadol Once A Day | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 9 | 1
Other Adverse Events (participants affected / at risk) | 136 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | 1 Tramadol Once A Day | 2 Placebo
Grand mal convulsion (Nervous system disorders) | 1/1023 (1) | 0/214 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1023 (1) | 0/214 (0)
Hepatitis (Infections and infestations) | 1/1023 (1) | 0/214 (0)
Renal impairment (Renal and urinary disorders) | 1/1023 (1) | 0/214 (0)
Popliteal bursitis (Musculoskeletal and connective tissue disorders) | 1/1023 (1) | 0/214 (0)
Ischaemic stroke (Nervous system disorders) | 0/1023 (0) | 1/214 (1)
Diverticulitis (Gastrointestinal disorders) | 1/1023 (1) | 0/214 (0)
Angina unstable (Cardiac disorders) | 1/1023 (1) | 0/214 (0)
Syncope (Nervous system disorders) | 1/1023 (1) | 0/214 (0)
Chest pain (General disorders) | 1/1023 (1) | 0/214 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1023 (1) | 0/214 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | 1 Tramadol Once A Day | 2 Placebo
Nausea (Gastrointestinal disorders) | 66/432 (86) | 12/214 (12)
Constipation (Gastrointestinal disorders) | 61/432 (73) | 9/214 (12)
Dizziness (Nervous system disorders) | 26/432 (28) | 7/214 (8)
Somnolence (Nervous system disorders) | 29/432 (40) | 8/214 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.